CLINICAL TRIAL: NCT05001854
Title: Evaluation of the Hemodynamics Effects of Fludrocortisone on the Pressor Response to Noradrenaline in Septic Shock Patients
Brief Title: Hemodynamics Effects of Fludrocortisone on the Pressor Response to Noradrenaline Septic Shock Patients
Acronym: FLUDROSEPSIS
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: study suspended until new therapeutic units are available
Sponsor: Rennes University Hospital (Other)
Collaborators: H.A.C. PHARMA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35RC19_8860; 2020-001430-35 (EudraCT Number)
Record Dates: First submitted 2021-07-08; First posted 2021-08-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Fludrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fludrocortisone (Experimental): 100 μg every 6 hours of fludrocortisone per os
  A pharmacokinetic study is performed in this arm
  Interventions: Drug: Fludrocortisone
- Control (Placebo Comparator): 100 μg every 6 hours of placebo per os
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fludrocortisone — 100 μg every 6 hours of fludrocortisone per os
  Other Names: Flucortac
  Arms: Fludrocortisone
Drug: Placebo — 100 μg every 6 hours of placebo per os
  Arms: Control

SUMMARY:
The benefit of low-dose steroids in septic shock is still debated today, especially with mineralocorticoids. Fludrocortisone is a synthetic mineralocorticoid, an analogue of aldosterone, which has shown, in combination with hydrocortisone, a favorable effect on the mortality of septic shock patients with relative adrenal insufficiency. In a previous study in healthy volunteers, we showed for the first time that fludrocortisone at a dose of 400 μg per day significantly improved the pressor response to phenylephrine. These results confirm the observations reported in rats with endotoxin shock, where fludrocortisone was shown to significantly increase blood pressure and contractile response to phenylephrine. These encouraging results argue for a potential vascular beneficial effect of fludrocortisone and need to be confirmed in a population of septic shock patients. In this context, we aimed to evaluate the effect of oral administration of 100 μg every 6 hours of fludrocortisone on vascular responsiveness to noradrenaline in septic shock patients.

DETAILED DESCRIPTION:
Patients admitted to medical and surgical intensive care units with septic shock who meet the selection criteria may be offered participation in the study. The consent is signed either by the patient or his or her relative/legal representative if he or she is not capable or the patient is included according to the emergency procedure in the absence of a relative. The patient is managed according to the usual procedures for patients in septic shock. After collection of the initial workup and basal measurements, the physician randomizes (=includes) the patient into one of 2 arms : the patient receives either fludrocortisone (400 μg per day), administered in 1 dose of 100 μg every 6 hours, i.e., 2 tablets of 50 μg per dose, or the placebo

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient with septic shock for less than 48 hours, defined by the combination of:

  * Sepsis defined as organ dysfunction caused by an inappropriate host response to infection (increase in SOFA score of at least 2 points secondary to infection),
  * Persistent hypotension requiring vasopressor drugs to maintain mean arterial pressure ≥ 65 mmHg,
* Hemodynamic stability for >30 min with mean arterial pressure ≥ 65 mmHg and noradrenaline dose ≤ 0.5 μg/kg/min,
* Consent signed by the patient, family member, or legal representative or inclusion under emergency procedure,
* Negative to a diagnostic test for SARS-CoV2 less than 72 hours old; the test used must be on the the list published on the Ministry of Solidarity and Health website

Non-inclusion Criteria:

* Current treatment with steroids or other treatment that may affect the hypothalamic-pituitary-adrenal axis,
* Anesthetic induction with etomidate within 6 hours prior to randomization given its selective inhibitory effect on 11 β-hydroxylase,
* Known hypersensitivity to fludrocortisone (or any of its excipients), or to tetracosactide (Synacthen®),
* Disturbed gastric emptying (gastric residue > 500 ml) in the absence of an alternative route of administration available (naso-jejunal tube or jejunostomy),
* Pregnant or nursing woman,
* Patient participating in another trial, possibly interfering with the study procedures,
* Person not affiliated to a social security system,
* Known situation of deprivation of freedom (safeguard of justice), guardianship or curatorship,
* Patient with a life expectancy of less than 24 hours.
* Patient with known or suspected SARS-CoV2 pneumonia

Exclusion criteria:

* Patients under court protection will be excluded as soon as the investigator is aware of their status.
* Hemodynamic worsening with noradrenaline dose >1.5 μg/kg/min before evaluation of the primary end point.
* Catecholamine withdrawal before evaluation of the primary end point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mean arterial blood pressure (mmHg) | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  Mean arterial blood pressure (mmHg) after a dose escalation of norepinephrine in increments of 0.2 μg/kg/min to a maximum dose of 1.5 μg/kg/min.

SECONDARY OUTCOMES:
Heart rate | Baseline, before the first administration of the drug (fludrocortisone/placebo)
  Heart rate
Heart rate | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  Heart rate
Heart rate | After the 3rd administration of fludrocortisone or placebo (12 hours)
  Heart rate
Heart rate | After the 4th administration of fludrocortisone or placebo (18 hours)
  Heart rate
arterial pressure | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  Mean arterial pressure, systolic arterial pressure, diasystolic arterial pressure
arterial pressure | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  Mean arterial pressure, systolic arterial pressure, diasystolic arterial pressure
arterial pressure | After the 3rd administration of fludrocortisone or placebo (12 hours)
  Mean arterial pressure, systolic arterial pressure, diasystolic arterial pressure
arterial pressure | After the 4th administration of fludrocortisone or placebo (18 hours)
  Mean arterial pressure, systolic arterial pressure, diasystolic arterial pressure
Cardiac output | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  Cardiac output
Cardiac output | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  Cardiac output
Cardiac output | After the 3rd administration of fludrocortisone or placebo (12 hours)
  Cardiac output
Cardiac output | After the 4th administration of fludrocortisone or placebo (18 hours)
  Cardiac output
Cardiac index | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  Cardiac index
Cardiac index | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  Cardiac index
Cardiac index | After the 3rd administration of fludrocortisone or placebo (12 hours)
  Cardiac index
Cardiac index | After the 4th administration of fludrocortisone or placebo (18 hours)
  Cardiac index
Indexed Systemic Vascular Resistances (ISVR) | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  Indexed Systemic Vascular Resistances (ISVR)
Indexed Systemic Vascular Resistances (ISVR) | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  Indexed Systemic Vascular Resistances (ISVR)
Indexed Systemic Vascular Resistances (ISVR) | After the 3rd administration of fludrocortisone or placebo (12 hours)
  Indexed Systemic Vascular Resistances (ISVR)
Indexed Systemic Vascular Resistances (ISVR) | After the 4th administration of fludrocortisone or placebo (18 hours)
  Indexed Systemic Vascular Resistances (ISVR)
Indexed Global Telediastolic Volume (IGVT) | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  Indexed Global Telediastolic Volume (IGVT)
Indexed Global Telediastolic Volume (IGVT) | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  Indexed Global Telediastolic Volume (IGVT)
Indexed Global Telediastolic Volume (IGVT) | After the 3rd administration of fludrocortisone or placebo (12 hours)
  Indexed Global Telediastolic Volume (IGVT)
Indexed Global Telediastolic Volume (IGVT) | After the 4th administration of fludrocortisone or placebo (18 hours)
  Indexed Global Telediastolic Volume (IGVT)
Ejection Volume Variability (EVV) | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  Ejection Volume Variability (EVV)
Ejection Volume Variability (EVV) | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  Ejection Volume Variability (EVV)
Ejection Volume Variability (EVV) | After the 3rd administration of fludrocortisone or placebo (12 hours)
  Ejection Volume Variability (EVV)
Ejection Volume Variability (EVV) | After the 4th administration of fludrocortisone or placebo (18 hours)
  v
Extravascular Pulmonary Water (EVW) | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  Extravascular Pulmonary Water (EVW)
Extravascular Pulmonary Water (EVW) | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  Extravascular Pulmonary Water (EVW)
Extravascular Pulmonary Water (EVW) | After the 3rd administration of fludrocortisone or placebo (12 hours)
  Extravascular Pulmonary Water (EVW)
Extravascular Pulmonary Water (EVW) | After the 4th administration of fludrocortisone or placebo (18 hours)
  Extravascular Pulmonary Water (EVW)
Mortality | Day 28
  Percentage of deceased patients
Mortality | Day 90
  Percentage of deceased patients
Length of stay in intensive care unit | Day 90
  Length of stay in intensive care unit
Length of stay in care unit | Day 90
  Length of stay in care unit
Time to wean from catecholamines | Day 90
  Time to wean from catecholamines
Duration of mechanical ventilation (MV) | Day 90
  Duration of mechanical ventilation (MV)
Inflammation markers | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  IFNγ, TNF α, IL1β, IL6, IL10 dosage
Inflammation markers | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  IFNγ, TNF α, IL1β, IL6, IL10 dosage
natremia dosage | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  blood sodium
natremia dosage | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  blood sodium
urinary sodium dosage | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  urinary sodium
urinary sodium dosage | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  urinary sodium
kalemia dosage | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  blood potassium
kalemia dosage | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  blood potassium
urinary potassium dosage | Baseline, before the first administration of the experimental drug (fludrocortisone/placebo)
  urinary potassium
urinary potassium dosage | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  urinary potassium
pharmacokinetics of fludrocortisone : Area under the plasma concentration-time curve (plasma concentrations of fludrocortisone at 5 times) | After 4th dose of fludrocortisone (18 hours)
  in the experimental group only.

OTHER OUTCOMES:
Dose-response relationship | 1,5 hours after the second administration of fludrocortisone or placebo (7,5 hours)
  The dose-response relationship (mean arterial blood pressure to doses of norepinephrine) will be modeled according to a sigmoid Emax model with determination of the maximum effect (Emax) obtained on blood pressure, estimation of the dose of norepinephrine inducing half of the Emax (ED50), and the Hill coefficient γ reflecting the sigmoidality of the curve.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Laviolle, MD, PhD, Study Chair — Rennes University Hospital; Harmonie Perrichet, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital - Intensive Care unit, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No